CLINICAL TRIAL: NCT00577122
Title: MPA Revisited: A Phase II Study of Anti-Metastatic, Anti-Angiogenic Therapy in Postmenopausal Patients With Hormone Receptor Negative Breast Cancer. A Translational Breast Cancer Research Consortium (TBCRC) Trial
Brief Title: Medroxyprogesterone +/- Cyclophosphamide & Methotrexate in Hormone Receptor-Negative Recurrent/Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Translational Breast Cancer Research Consortium (Other)
Responsible Party: Principal Investigator, Kathy Miller, Ballvé-Lantero Professor of Medicine, Indiana University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0607-18 IUCRO-0154; TBCRC 007 (Other: Translational Breast Cancer Reserach Consortium)
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Results first posted 2014-09-23 (Estimated); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Estrogen Receptor-negative Breast Cancer; Progesterone Receptor-negative Breast Cancer; Recurrent Breast Cancer; Stage IV Breast Cancer
Keywords: Medroxyprogesterone progesterone acetate (MPA); Cyclophosphamide plus Methotrexate
MeSH Terms: conditions — Breast Neoplasms | interventions — Medroxyprogesterone; Medroxyprogesterone Acetate; Cyclophosphamide; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort I (MPA) (Experimental): Medroxyprogesterone progesterone acetate (MPA) will be administered orally as a single daily dose.
  Interventions: Drug: Medroxyprogesterone progesterone acetate (MPA)
- Cohort II (MPA, low-dose chemotherapy) (Experimental): Medroxyprogesterone progesterone acetate (MPA) will be administered orally as a single daily dose.
  Cyclophosphamide will be administered orally as a single daily dose. Methotrexate will be administered twice daily on days 1 and 2 of each week.
  Interventions: Drug: Medroxyprogesterone with Cyclophosphamide + Methotrexate

INTERVENTIONS:
Drug: Medroxyprogesterone progesterone acetate (MPA) — 1000 mg po daily
  Other Names: (6alpha)-17-hydroxy-6-methylpregn-4-ene-3,20-dione; 17alpha-hydroxy-6alpha-methylprogesterone; 27408; 520-85-4; 6alpha-methyl-17alpha-hydroxyprogesterone; 6alpha-methyl-4-pregnen-17alpha-ol-3,20-dione; Curretab; Depo-Provera; Provera; Provera Dosepak
  Arms: Cohort I (MPA)
Drug: Medroxyprogesterone with Cyclophosphamide + Methotrexate — Medroxyprogesterone Acetate Dose 1000 mg po daily Cyclophosphamide Dose 50 mg po daily Methotrexate Dose 2.5 mg po daily Days 1 and 2 of each week
  Other Names: medroxyprogesterone acetate; MPA; cyclophosphamid monohydrate; CTX; methylaminopterin; MTX
  Arms: Cohort II (MPA, low-dose chemotherapy)

SUMMARY:
The purpose of this study is to evaluate the impact of MPA alone and in combination with low dose oral chemotherapy in patients with ER- and PR- advanced breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the clinical benefit rate (complete response [CR] + partial response [PR] + stable disease [SD] >= 6 months) of medroxyprogesterone acetate (MPA) monotherapy and MPA + low dose oral cyclophosphamide and methotrexate (ldoCM) in patients with refractory hormone receptor negative metastatic breast cancer.

SECONDARY OBJECTIVES:

I. To evaluate the toxicity of MPA and MPA + ldoCM in this patient population. II. To explore the relationship between MPA trough level and clinical benefit. III. To explore genetic determinants of MPA bioavailability and trough concentration.

IV. To explore potential surrogates of biologic activity including Nm-23 expression in primary tumor, change in Nm-23 expression in skin, change in plasma thrombospondin (TSP)-1, change in plasma plasminogen activator inhibitor (PAI)-1 antigen and activity.

OUTLINE: Patients are assigned to 1 of 2 treatment arms.

COHORT I: Patients receive MPA orally (PO) once daily (QD).

COHORT II: Patients receive MPA as in Cohort I, cyclophosphamide PO QD, and methotrexate PO twice daily (BID) on days 1 and 2 of every week.

In both arms, treatment continues in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the breast with measurable locally recurrent or metastatic disease
* Primary tumor must be ER negative and PR negative
* Patients must be post-menopausal
* Patients may have had up to 3 prior chemotherapy regimens for recurrent/metastatic disease
* Adequate organ function as evidenced by laboratory studies outlined in section 3.6 of the protocol
* Patients with treated, asymptomatic brain metastases are eligible provided chronic steroid therapy is not required

Exclusion Criteria:

* Patients must not have extensive pleural effusion or ascites
* Patients must not have history of DVT or pulmonary embolism w/in past 12 mo
* Patients must not have had chemotherapy or hormonal therapy within 2 weeks of study entry
* Patients must not have had radiation therapy within 1 week of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Miller, MD, Principal Investigator — IU Simon Cancer Center
Locations (7):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, San Francisco Comprehensive Cancer Center, San Francisco, California
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of North Carolina, Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Comprehensive Cancer Center, Durham, North Carolina
  - The University of Texas M. D. Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Since there was not enough evidence of clinical benefit, this study did not go beyond the first stage in the two stage design. A total of 30 patients (14 in the MPA alone cohort and 16 in the MPA+ ldoCM cohort) were in the study before the study ended.
Groups:
- Cohort 1: MPA-Alone: Medroxyprogesterone progesterone acetate (MPA) will be administered orally as a single daily dose.
- Cohort 2: MPA+IdoCM: Medroxyprogesterone progesterone acetate (MPA) will be administered orally as a single daily dose.
  Cyclophosphamide will be administered orally as a single daily dose. Methotrexate will be administered twice daily on days 1 and 2 of each week.
Period: Overall Study
Arm/Group | Cohort 1: MPA-Alone | Cohort 2: MPA+IdoCM
Started | 14 | 16
Completed | 0 | 0
Not Completed | 14 | 16
Not completed — Adverse Event | 0 | 2
Not completed — Progression, relapse during active trt | 6 | 8
Not completed — Prog, refract disease during active trt | 8 | 5
Not completed — Alternative Therapy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: MPA-Alone | Cohort 2: MPA+IdoCM | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 12 | 21
  >=65 years | 5 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.0 (12.78) | 56.2 (12.24) | 57.5 (12.36) [0 to 0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 16 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 9 | 12 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate (CR + PR + SD > 6 Months).
Description: To determine the clinical benefit rate (Complete Response + Partial Response + Stable Disease > 6 months) per Response Evaluation Criteria in Solid tumors (RECIST version 1.0). of MPA monotherapy and MPA + low dose oral cyclophosphamide and methotrexate (ldoCM) in patients with refractory hormone receptor negative metastatic breast cancer. This will show the percent of patients who had Clinical Benefit and the Exact 95% Confidence Interval.
Time Frame: baseline through end of study, up to 3 years
Population: All Patients on study.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Groups:
- Cohort I: MPA-Alone: Medroxyprogesterone progesterone acetate (MPA) will be administered orally as a single daily dose.
Arm/Group | Cohort I: MPA-Alone | Cohort 2: MPA+IdoCM
Number analyzed (Participants) | 14 | 16
Percent of Participants | 7.1 [0.2 to 33.9] | 6.3 [0.2 to 30.2]

2. Secondary Outcome: Grade 3 or 4 Adverse Events Related to Treatment
Description: To evaluate the toxicity of MPA and MPA + ldoCM in this patient population by the number of patients who have grade 3 or 4 adverse events that are related to treatment.
Time Frame: baseline through end of treatment
Population: All patients in the study
Measure: Number; unit: participants
Groups:
- Cohort II: MPA+IdoCM: Medroxyprogesterone progesterone acetate (MPA) will be administered orally as a single daily dose.
  Cyclophosphamide will be administered orally as a single daily dose. Methotrexate will be administered twice daily on days 1 and 2 of each week.
Arm/Group | Cohort I: MPA-Alone | Cohort II: MPA+IdoCM
Number analyzed (Participants) | 14 | 16
participants | 2 | 2

3. Secondary Outcome: MPA Trough Level > 50 ng/mL When Have Clinical Benefit
Description: To explore the relationship between MPA trough level and clinical benefit. This is done by seeing if the MPA concentrations remained > 50 ng/mL after initial dose escalation for those patients who showed clinical benefit. The number shows how many of the patients who showed clinical benefit had MPA concentrations > 50 ng/mL.
Time Frame: baseline through end of treatment
Population: Patients who showed clinical benefit (CR, PR, or SD > 6 months)
Measure: Number; unit: participants
Arm/Group | Cohort I: MPA-Alone | Cohort II: MPA+IdoCM
Number analyzed (Participants) | 1 | 1
participants | 1 | 1

4. Secondary Outcome: MPA Trough Concentration
Description: To explore genetic determinants of MPA bioavailability and trough concentration by showing average MPA levels at cycle 1 (Day 10-14) and cycle 2 (Day 1).
Time Frame: Cycle 1 (Day 10-14) and Cycle 2 (Day 1)
Population: All patients with available data
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort I: MPA-Alone | Cohort II: MPA+IdoCM
Number analyzed (Participants) | 14 | 16
ng/mL
  Cycle 1, Day 10-14 | 14.5 (8.9) | 42.1 (66.4)
  Cycle 2, Day 1 | 52.6 (65.3) | 66.4 (71.5)

ADVERSE EVENTS:
Time Frame: Throughout the entire study, up to 3 years.
Groups:
- Cohort 1: MPA Alone: Medroxyprogesterone progesterone acetate (MPA) will be administered orally as a single daily dose.
Arm/Group | Cohort 1: MPA Alone | Cohort 2: MPA+IdoCM
Serious Adverse Events (participants affected / at risk) | 2/14 | 2/16
Other Adverse Events (participants affected / at risk) | 14/14 | 12/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: MPA Alone (N=14) | Cohort 2: MPA+IdoCM (N=16)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
FRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 1 (1)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: MPA Alone (N=14) | Cohort 2: MPA+IdoCM (N=16)
DERMAL CHANGE LYMPHEDEMA, PHLEBOLYMPHEDEMA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
LYMPHATICS (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
AUDITORY/EAR (Ear and labyrinth disorders) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 5 (5) | 4 (4)
DIARRHEA (Gastrointestinal disorders) | 1 (1) | 2 (2)
DRY MOUTH/SALIVARY GLAND (XEROSTOMIA) (Gastrointestinal disorders) | 1 (1) | 0 (0)
DYSPHAGIA (DIFFICULTY SWALLOWING) (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRITIS (INCLUDING BILE REFLUX GASTRITIS) (Gastrointestinal disorders) | 1 (1) | 1 (1)
GASTROINTESTINAL - OTHER (SPECIFY, __) (Gastrointestinal disorders) | 0 (0) | 2 (2)
HEARTBURN/DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 1 (1)
MUCOSITIS/STOMATITIS (CLINICAL EXAM) - STOMACH (Gastrointestinal disorders) | 0 (0) | 1 (1)
MUCOSITIS/STOMATITIS (FUNCTIONAL/SYMPTOMATIC) - ESOPHAGUS (Gastrointestinal disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 3 (3) | 3 (3)
PAIN - ABDOMEN NOS (Gastrointestinal disorders) | 0 (0) | 2 (2)
TASTE ALTERATION (DYSGEUSIA) (Gastrointestinal disorders) | 3 (3) | 1 (1)
VOMITING (Gastrointestinal disorders) | 2 (2) | 0 (0)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 7 (7) | 7 (7)
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 0 (0) | 2 (2)
PAIN - OTHER (SPECIFY, __) (General disorders) | 3 (3) | 3 (3)
INFECTION - OTHER (SPECIFY, __) (Infections and infestations) | 0 (0) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - BLADDER (URINARY) (Infections and infestations) | 0 (0) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - LUNG (PNEUMONIA) (Infections and infestations) | 0 (0) | 1 (1)
INFECTION WITH UNKNOWN ANC - NECK NOS (Infections and infestations) | 1 (1) | 0 (0)
PAIN - SKIN (Infections and infestations) | 0 (0) | 1 (1)
BURN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ALKALINE PHOSPHATASE (Investigations) | 0 (0) | 1 (1)
ALT, SGPT (SERUM GLUTAMIC PYRUVIC TRANSAMINASE) (Investigations) | 0 (0) | 1 (1)
AST, SGOT(SERUM GLUTAMIC OXALOACETIC TRANSAMINASE) (Investigations) | 1 (1) | 0 (0)
BICARBONATE, SERUM-LOW (Investigations) | 1 (1) | 0 (0)
HEMOGLOBIN (Investigations) | 2 (2) | 0 (0)
INR (INTERNATIONAL NORMALIZED RATIO OF PROTHROMBIN TIME) (Investigations) | 2 (2) | 0 (0)
METABOLIC/LABORATORY - OTHER (SPECIFY, __) (Investigations) | 0 (0) | 1 (1)
PTT (PARTIAL THROMBOPLASTIN TIME) (Investigations) | 1 (1) | 0 (0)
WEIGHT GAIN (Investigations) | 0 (0) | 1 (1)
ANOREXIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
CALCIUM, SERUM-LOW (HYPOCALCEMIA) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
POTASSIUM, SERUM-LOW (HYPOKALEMIA) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
URIC ACID, SERUM-HIGH (HYPERURICEMIA) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
EDEMA: LIMB (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
PAIN - BACK (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
PAIN - BONE (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
PAIN - CHEST WALL (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
PAIN - CHEST/THORAX NOS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
PAIN - EXTREMITY-LIMB (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
PAIN - JOINT (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
PAIN - MUSCLE (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
PAIN - NECK (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN - PAIN NOS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 0 (0)
NEUROLOGY - OTHER (SPECIFY, __) (Nervous system disorders) | 0 (0) | 1 (1)
NEUROPATHY: SENSORY (Nervous system disorders) | 6 (6) | 2 (2)
PAIN - HEAD/HEADACHE (Nervous system disorders) | 1 (1) | 2 (2)
PAIN - NEURALGIA/PERIPHERAL NERVE (Nervous system disorders) | 0 (0) | 1 (1)
SPEECH IMPAIRMENT (E.G., DYSPHASIA OR APHASIA) (Nervous system disorders) | 1 (1) | 0 (0)
SWEATING (DIAPHORESIS) (Nervous system disorders) | 2 (2) | 0 (0)
TREMOR (Nervous system disorders) | 1 (1) | 0 (0)
INSOMNIA (Psychiatric disorders) | 5 (5) | 5 (5)
MOOD ALTERATION - AGITATION (Psychiatric disorders) | 0 (0) | 1 (1)
MOOD ALTERATION - ANXIETY (Psychiatric disorders) | 4 (4) | 2 (2)
MOOD ALTERATION - DEPRESSION (Psychiatric disorders) | 4 (4) | 2 (2)
HOT FLASHES/FLUSHES (Reproductive system and breast disorders) | 4 (4) | 2 (2)
IRREGULAR MENSES (CHANGE FROM BASELINE) (Reproductive system and breast disorders) | 0 (0) | 1 (1)
MEMORY IMPAIRMENT (Reproductive system and breast disorders) | 1 (1) | 1 (1)
PAIN - BREAST (Reproductive system and breast disorders) | 2 (2) | 1 (1)
VAGINAL DRYNESS (Reproductive system and breast disorders) | 0 (0) | 1 (1)
ALLERGIC RHINITIS (INCLUDING SNEEZING, NASAL STUFFINESS, POSTNASAL DRIP) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5)
DIZZINESS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (7)
HICCOUGHS (HICCUPS, SINGULTUS) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
NASAL CAVITY/PARANASAL SINUS REACTIONS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
VOICE CHANGES/DYSARTHRIA (E.G., HOARSENESS, LOSS OR ALTERATION IN VOICE, LARYNGITIS) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
ATROPHY, SKIN (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DERMATOLOGY/SKIN - OTHER (SPECIFY, __) (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
HAIR LOSS/ALOPECIA (SCALP OR BODY) (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
MUCOSITIS/STOMATITIS (CLINICAL EXAM) - ORAL CAVITY (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
NAIL CHANGES (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
ULCERATION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes